CLINICAL TRIAL: NCT04789889
Title: Comparison of Satisfaction With Conserved Breast, Postoperative Complications and Tumor Control Between IORT and Postoperative Radiotherapy in Breast Conserving Surgery
Brief Title: Comparison Between IORT and Postoperative Radiotherapy in Breast Conserving Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The intraoperative radiotherapy machine was out of order and could not be used.
Sponsor: Xiangyun Zong (Other)
Responsible Party: Sponsor-Investigator, Xiangyun Zong, Director of Breast Cancer, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Organization: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JTU-6H-20210227001
Record Dates: First submitted 2021-03-02; First posted 2021-03-10 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2023-01

CONDITIONS: Quality of Life
Keywords: intraoperative radiotherapy; breast-conserving surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IORT (Experimental): intraoperative radiotherapy(IORT) in BCS.
  Interventions: Radiation: intraoperative radiotherapy
- PORT (Active Comparator): traditional postoperative radiotherapy following BCS.
  Interventions: Radiation: postoperative radiotherapy

INTERVENTIONS:
Radiation: intraoperative radiotherapy — intraoperative radiotherapy
  Arms: IORT
Radiation: postoperative radiotherapy — postoperative radiotherapy
  Arms: PORT

SUMMARY:
To compare the satisfaction with conserved breast, acute and chronic postoperative complications and tumor control between intraoperative radiotherapy(IORT) and traditional postoperative radiotherapy following breast-conserving surgery (BCS).

ELIGIBILITY:
Inclusion Criteria:

* Primary invasive breast cancer confirmed by pathology.
* Maximum tumor diameter ≤3.5cm.
* Clinical lymph nodes are negative.
* Single or multiple tumors are located on the same side of the nipple and in the same quadrant.
* ECOG status score ≤ 2.
* With informed Consents.

Exclusion Criteria:

* Previous history of breast cancer or other malignant tumors.
* Inflammatory breast cancer; 3. Previous radiotherapy history.
* Other diseases affecting radiotherapy, such as connective tissue disease, heart disease, lung disease and so on.
* Patients who are not going to have the axillary lymph node surgery (including SLN and ALND) were excluded.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Rate of successful surgical procedure | immediately after surgery
  the rate of successful breast conserving surgery
satisfaction with conserved breast | 1 month after surgery
  the patients' satisfaction to postoperative breast including shape and feeling(Harvard/NSABP/RTOG BREAST COSMETIC SCALE: excellent, good, fair, poor)

SECONDARY OUTCOMES:
Rate of acute and chronic postoperative complications（CTCAE 3.0) | 1-month, 6-month after surgery
  The incidence of adverse reactions at 1 and 6 months after operation
DFS | 2-3 years after surgery
  long-term postoperative disease-free survival
OS | 2-3 years after surgery
  long-term postoperative overall survival

CONTACTS AND LOCATIONS:
Overall Officials: ZONG, MD, PhD, Study Director — Shanghai Jiao Tong University affiliated 6th Hospital
Locations (1):
- Shanghai Jiao Tong University Affiliated Sixth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kawamura M, Itoh Y, Kamomae T, Sawaki M, Kikumori T, Tsunoda N, Ito J, Shimoyama Y, Satake H, Naganawa S. A phase I/II trial of intraoperative breast radiotherapy in an Asian population: 10-year results with critical evaluation. J Radiat Res. 2020 Jul 6;61(4):602-607. doi: 10.1093/jrr/rraa029. PMID 32494808
- [Background] Wang L, Zhu M, Cui Y, Zhang X, Li G. Efficacy analysis of intraoperative radiotherapy in patients with early-stage breast cancer. Cancer Cell Int. 2020 Sep 11;20:446. doi: 10.1186/s12935-020-01533-z. eCollection 2020. PMID 32943994
- [Background] Forster T, Jakel C, Akbaba S, Krug D, Krempien R, Uhl M, Hafner MF, Konig L, Koerber SA, Harrabi S, Bernhardt D, Behnisch R, Krisam J, Hennigs A, Sohn C, Heil J, Debus J, Horner-Rieber J. Fatigue following radiotherapy of low-risk early breast cancer - a randomized controlled trial of intraoperative electron radiotherapy versus standard hypofractionated whole-breast radiotherapy: the COSMOPOLITAN trial (NCT03838419). Radiat Oncol. 2020 Jun 1;15(1):134. doi: 10.1186/s13014-020-01581-9. PMID 32487184
- [Background] Hu X, He Y, Chen X, Xia T, Cao T, Jia H, Zhang L. Impact of intraoperative radiotherapy on the perioperative period of patients after breast-conserving surgery. Gland Surg. 2020 Oct;9(5):1535-1542. doi: 10.21037/gs-20-727. PMID 33224829
- [Background] Gondim GRM, Makdissi FBA, Fogaroli RC, Collins JBD, Iyeyasu H, de Castro DG, Silva MLG, Chen MJ, Coelho TM, Ramos H, Pellizzon ACA. Intraoperative breast radiotherapy: survival, local control and risk factors for recurrence. Rep Pract Oncol Radiother. 2019 Nov-Dec;24(6):551-555. doi: 10.1016/j.rpor.2019.09.004. Epub 2019 Oct 16. PMID 31660047
- [Background] Uhlig S, Wuhrer A, Berlit S, Tuschy B, Sutterlin M, Bieback K. Intraoperative radiotherapy for breast cancer treatment efficiently targets the tumor bed preventing breast adipose stromal cell outgrowth. Strahlenther Onkol. 2020 Apr;196(4):398-404. doi: 10.1007/s00066-020-01586-z. Epub 2020 Feb 6. PMID 32030446
- [Background] Sasieni PD, Sawyer EJ. Intraoperative radiotherapy for early breast cancer - insufficient evidence to change practice. Nat Rev Clin Oncol. 2020 Dec;17(12):723-724. doi: 10.1038/s41571-020-00444-2. PMID 33087894
- [Background] Vaidya JS, Bulsara M, Baum M, Alvarado M, Bernstein M, Massarut S, Saunders C, Sperk E, Wenz F, Tobias JS; TARGIT-A investigators. Intraoperative radiotherapy for breast cancer: powerful evidence to change practice. Nat Rev Clin Oncol. 2021 Mar;18(3):187-188. doi: 10.1038/s41571-021-00471-7. No abstract available. PMID 33495552
- [Background] Vaidya JS, Bulsara M, Baum M, Wenz F, Massarut S, Pigorsch S, Alvarado M, Douek M, Saunders C, Flyger HL, Eiermann W, Brew-Graves C, Williams NR, Potyka I, Roberts N, Bernstein M, Brown D, Sperk E, Laws S, Sutterlin M, Corica T, Lundgren S, Holmes D, Vinante L, Bozza F, Pazos M, Le Blanc-Onfroy M, Gruber G, Polkowski W, Dedes KJ, Niewald M, Blohmer J, McCready D, Hoefer R, Kelemen P, Petralia G, Falzon M, Joseph DJ, Tobias JS. Long term survival and local control outcomes from single dose targeted intraoperative radiotherapy during lumpectomy (TARGIT-IORT) for early breast cancer: TARGIT-A randomised clinical trial. BMJ. 2020 Aug 19;370:m2836. doi: 10.1136/bmj.m2836. PMID 32816842
- [Background] Onthong K, Chakkabat C, Nantavithya C, Shotelersuk K, Denariyakoon S, Vongsaisuwon M, Chulakadabbav A, Chatamra K, Saksornchai K. Results of intraoperative radiotherapy given as a boost after breast conserving-surgery. Gland Surg. 2020 Oct;9(5):1389-1395. doi: 10.21037/gs-20-249. PMID 33224814
- [Background] Vaidya JS, Bulsara M, Baum M, Tobias JS; TARGIT-A trial authors. Single-dose intraoperative radiotherapy during lumpectomy for breast cancer: an innovative patient-centred treatment. Br J Cancer. 2021 Apr;124(9):1469-1474. doi: 10.1038/s41416-020-01233-5. Epub 2021 Feb 2. PMID 33531693
- [Background] Feng K, Meng X, Liu J, Xing Z, Zhang M, Wang X, Feng Q, Wang X. Update on intraoperative radiotherapy for early-stage breast cancer. Am J Cancer Res. 2020 Jul 1;10(7):2032-2042. eCollection 2020. PMID 32774999